CLINICAL TRIAL: NCT05142800
Title: Screening for Edema and Breast Cancer-Related Lymphedema in Patients Undergoing Targeted Therapy for Breast Cancer
Brief Title: Screening For BCRL In Targeted Therapy For Breast Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Heinz Family Foundation (Unknown)
Responsible Party: Principal Investigator, Alphonse Taghian, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 18-195
Record Dates: First submitted 2021-11-15; First posted 2021-12-03 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Lymphedema; Lymphedema Arm; Lymphedema of Upper Arm; Lymphedema of Upper Limb; Lymphedema of the Hands; Edema; Edema Arm; Breast Cancer Lymphedema; Breast Cancer Metastatic; Breast Cancer Stage; Breast Cancer
Keywords: Lymphedema; Lymphedema Arm; Lymphedema of Upper Arm; Lymphedema of Upper Limb; Lymphedema of the Hands; Edema; Edema Arm; Breast Cancer Lymphedema; Breast Cancer Metastatic; Breast Cancer Stage; Breast Cancer
MeSH Terms: conditions — Lymphedema; Edema; Breast Cancer Lymphedema; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Target Therapy Drug-Stand Care: Screening procedures confirm participation in the research study.
  * Participants limb volume is measured prior to treatment start date.
  * Participant is provided informational brochure about risk of lymphedema and Lymphedema Screening Program Card.
  * Perometer and SOZO measurements will be incorporated as a part of the follow-up visits throughout the course of their trial and for at least 6 months beyond their last dose of trial medication
  Interventions: Device: Perometer; Device: SOZO device
- Target Therapy-Early or Metastatic Breast Cancer: Screening procedures confirm participation in the research study.
  * Participants limb volume is measured prior to treatment start date.
  * Participant is provided informational brochure about risk of lymphedema and Lymphedema Screening Program Card.
  * Perometer and SOZO measurements will be incorporated as a part of the follow-up visits throughout the course of their trial and for at least 6 months beyond their last dose of trial medication
  Interventions: Device: Perometer; Device: SOZO device

INTERVENTIONS:
Device: Perometer — The perometer uses light sensors to calculate the length and volume of your arms
Device: SOZO device — The machine measures the amount of fluid on the arm(s)

SUMMARY:
This a prospective, longitudinal study designed to track edema and Breast Cancer Related Lymphedema (BCRL) onset in breast cancer patients taking targeted therapy treatments for early and metastatic breast cancer.

A Perometer and Sozo devise will be used to measure volume changes

DETAILED DESCRIPTION:
This study will compare patients' relative arm volume changes and symptoms data from before drug therapy throughout drug treatment and for up to six months after treatment has finished.

A Perometer and Sozo device will be used to measure volume changes

All participants will be accrued at Massachusetts General Hospital for a target accrual of 166 participants.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are receiving treatment in the MGH Breast Cancer Center who are enrolled in a DF/HCC-regulated targeted therapy trial for the treatment of early or metastatic breast cancer or patients being treated with a targeted therapy that may alter their risk of developing edema or BCRL will be eligible.
* Subjects that will be eligible for the study include:
* Females between 18 and 80 years of age
* With a history of breast cancer
* 4 weeks or more post-surgery
* With or without edema
* Undergoing treatment with targeted therapy for early or metastatic disease.

Exclusion Criteria:

- Patients who cannot attain 90 degrees of shoulder abduction (position of measurement with Perometer).

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are receiving treatment in the MGH Breast Cancer Center who are enrolled in a DF/HCC-regulated targeted therapy trial for the treatment of early or metastatic breast cancer or patients being treated with a targeted therapy that may alter their risk of developing edema or BCRL will be eligible.
Sampling Method: Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with a greater than or equal to 10% arm volume change from the first pre-treatment (targeted therapy) measurement, detected by perometry, occurring at least three months after breast surgery | At least three months post surgery up to 5 years, assessed every 3 months
  Greater than or equal to 10% arm volume change from the first pre-treatment (targeted therapy) measurement, detected by perometry, occurring at least three months after breast surgery

SECONDARY OUTCOMES:
To assess the time course to lymphedema onset | 5 Years
  We will also attempt to look at any time course differences of lymphedema onset by plotting cumulative incidence curves of the study and control groups and comparing hazard rates after accounting for important covariates in a multivariate Cox proportional-hazards model.
To asses the correlation of different targeted therapies with lymphedema onset | 5 Years
  We will compare the incidence of lymphedema by type of targeted therapy drug (CDK4/6, PI3K, mTOR, AKT).

CONTACTS AND LOCATIONS:
Overall Officials: Alphonse G. Taghian, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation